CLINICAL TRIAL: NCT00775021
Title: A Clinical Comparison of Two Daily Disposable Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0814; ID08-34
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A/nelfilcon A (Active Comparator): etafilcon A contact lens worn first and nelfilcon A contact lens worn second
  Interventions: Device: etafilcon A; Device: nelfilcon A
- nelfilcon A/etafilcon A (Active Comparator): nelfilcon A contact lens worn first and etafilcon A contact lens second.
  Interventions: Device: etafilcon A; Device: nelfilcon A

INTERVENTIONS:
Device: etafilcon A — Contact Lens
Device: nelfilcon A — Contact Lens

SUMMARY:
The objective of this study is to evaluate the clinical performance of two daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years to 45 years
* Current daily soft contact lens as habitual optical correction:
* Refraction:

  * Best sphere (corrected for back vertex distance) -1.00 to -6.00D
  * Cylinder 0.00 to - 0.75D
* Best spectacle corrected visual acuity of 6/9 or better in each eye
* Willingness to adhere to the instructions set in the clinical protocol
* Signature of the subject on the informed consent form

Exclusion Criteria:

* Systemic or ocular allergies which might interfere with contact lens wear
* Systemic disease which might interfere with contact lens wear
* Ocular disease which might interfere with contact lens wear (e.g. hypoesthesia, insufficient lacrimal secretion)
* Use of medication which might interfere with contact lens wear
* Active ocular infection
* Use of ocular medication
* Significant ocular anomaly
* Presence of two or more corneal scars in either eye
* Pregnancy or lactation
* Any medical condition that might be prejudicial to the study
* Participated in any other clinical studies in the past month
* Currently wears monovision

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Otometry Technology Group, Ltd., London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Etafilcon A/Nelfilcon A | Nelfilcon A/Etafilcon A
Started | 63 | 60
Completed | 62 | 60
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention
Arm/Group | Etafilcon A/Nelfilcon A | Nelfilcon A/Etafilcon A
Started | 62 | 60
Completed | 62 | 59
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Participants: Total number of participants that completed the study.
Arm/Group | Total Participants
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 41
Region of Enrollment [Number; unit: participants]
  United Kingdom | 121

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Subjects rated study contact lens for overall comfort using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 1 week
Population: Analysis includes all participants that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Etafilcon A: All subjects that wore etafilcon A contact lenses and completed the study.
- Nelfilcon A: All subjects that wore nelfilcon A contact lenses and completed the study.
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 121 | 121
units on a scale | 3.6685 (0.1141) | 3.4352 (0.1148)
Statistical Analysis 1: Comparison: Etafilcon A; The alternative hypothesis is that etafilcon A contact lenses will have equal to ro higher ratings of overall comfort than nelfilcon A contact lenses; Test type: Non-Inferiority or Equivalence — Margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = 0.2334, 95% CI 2-sided [-0.03501 to 0.2334], Standard Error of Mean 0.1618 — The mean difference is calculated as etafilconA minus nelfilcon A. Analysis is adjusted for lens type, period, lens type by period interaction, gender, lens type by gender interaction as fixed effects, subject nested within site as random effect

2. Secondary Outcome: Inferior Region Corneal Staining
Description: The investigator assessed abrasion to the lower portion of the cornea using the following scale:0 = None 1 = Slight micropunctate (1-10 spots) 2 = Moderate micropunctate (11-20 spots) 3 = Severe micropunctate (>20 spots)4 = Slight macropunctate (1-5 spots) 5 = Moderate macropuntate (>5-10 spots) 6 = Severe macropunctate (>10 spots) 7 = Slight patch (1-2mm)8 = Moderate patch (>2-4mm) 9 = Severe patch (>4mm)
Time Frame: 1 week
Population: Analysis includes all participants that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 121 | 121
units on a scale | 0.7004 (0.0643) | 0.8085 (0.0643)
Statistical Analysis 1: Comparison: Etafilcon A; The alternative hypothesis is that eyes that wore etafilcon A contact lenses will have less inferior region corneal staining than eyes that wore nelfilcon A contact lenses; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.1080, 98.7% CI 2-sided [-0.1080 to 0.06501], Standard Error of Mean 0.07768 — Mean difference calculated etafilcon A minus nelfilcon A. Analysis adjusted for lens type, period, lens by period interaction, gender, lens by gender interaction as fixed effects, subject nested within site and eye within subject as random effect

3. Secondary Outcome: End of the Day Comfort
Description: Subjects rated study contact lens comfort at the end of a day of lens wear using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 1 week
Population: Analysis includes all participants that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 121 | 121
units on a scale | 3.148 (0.127) | 2.7479 (0.1274)
Statistical Analysis 1: Comparison: Etafilcon A vs Nelfilcon A; The alternative hypothesis is that etafilcon A contact lenses have equal to or higher comfort ratings at the end of the day than nelfilcon A; Test type: Non-Inferiority or Equivalence — Margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = 0.4001, 98.7% CI 2-sided [-0.0055 to 0.4001], Standard Error of Mean 0.1799 — The mean difference is calculated as etafilcon A minus nelfilcon A

4. Secondary Outcome: Initial Comfort
Description: Subjects rated study contact lens for comfort immediately when they first put the lenses on using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 1 Week
Population: Analysis includes all participants that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 121 | 121
units on a scale | 3.5694 (0.1229) | 3.6783 (0.1233)
Statistical Analysis 1: Comparison: Etafilcon A vs Nelfilcon A; The alternative hypothesis is that etafilcon A contact lenses will have equal or higher ratings of initial comfort than nelfilcon A contact lenses; Test type: Non-Inferiority or Equivalence — Margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.1088, 98.7% CI 2-sided [-0.5016 to -0.1088], Standard Error of Mean 0.1741 — The mean difference is calculated as etafilcon A minus nelfilcon A

5. Secondary Outcome: Overall Lens Handling
Description: Subjects rated study contact lens for overall ease of handling using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 1 week
Population: Analysis includes all participants that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 121 | 121
units on a scale | 3.546 (0.1189) | 3.2971 (0.1187)
Statistical Analysis 1: Comparison: Etafilcon A vs Nelfilcon A; The alternative hypothesis is that etaflicon A contact lenses have equal to or higher ratings of ease of handling than nelfilcon A contact lenses; Test type: Non-Inferiority or Equivalence — Margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = 0.2489, 98.7% CI 2-sided [-0.1301 to 0.2489], Standard Error of Mean 0.168 — The mean difference is calculated as etafilcon A minus nelfilcon A

ADVERSE EVENTS:
Groups:
- Etafilcon A: etafilcon A contact lenses
- Nelfilcon A: nelfilcon A contact lenses.
Arm/Group | Etafilcon A | Nelfilcon A
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/122
Other Adverse Events (participants affected / at risk) | 0/122 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.